CLINICAL TRIAL: NCT04235829
Title: Predicting Weight Loss and Comorbid Improvement Early Post-operative Weight Loss Fails to Predict Outcomes 7 Years Following Laparoscopic Sleeve Gastrectomy: Does Early Weight Loss Matter
Brief Title: Does Early Weight Loss Following Laparoscopic Sleeve Gastrectomy Affect Long-term Outcomes
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, James Tankel, Resident in General Surgery, Shaare Zedek Medical Center
Other Study IDs: SZMC-95/19
Record Dates: First submitted 2019-11-30; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2; Gastrostomy; Morbid Obesity; Weight Loss
Keywords: sleeve gastrectomy; morbid obesity; predicting outcomes; early weight loss; hypertension; diabetes mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Obesity, Morbid; Weight Loss; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Form of obesity surgery

SUMMARY:
A study to explore the relationship between early weight loss in the 4 weeks following laparoscopic sleeve gastrectomy and outcomes, in terms of weight loss and comorbidity improvement, 7 years following the surgery.

DETAILED DESCRIPTION:
Patients who underwent laparoscopic sleeve gastrectomy in the 6 month period between 01/04/2012 and 01/10/2019 were identified. For those meeting the inclusion criteria, demographic and medical data was extracted from hospital notes. This included initial BMI and the presence of, or treatment for, diabetes or hypertension.

Using the contact details available in the medical records, a scripted telephone interview was performed. The current weight of the patient as well as a current medical and drug history were elicited. This data was compared with data attained during initial patient interaction with the service.

Early weight loss, defined as weight lost in the 4 weeks following surgery, was subsequently correlated with outcomes in terms of weight loss and improvement/resolution of either hypertension or diabetes at a 7 year follow up interval.

ELIGIBILITY:
Inclusion Criteria:

* LSG performed must have been the first surgical procedure performed for that the patient had undergone to treat their obesity
* Have not undergone any further bariatric surgical procedures since the index operation
* Still be alive at the time of the study
* Have correct be contactable with the contact details present available in the electronic database

Exclusion Criteria:

* Missing data
* Uncontactable
* Unwilling to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing laparoscopic sleeve gastrectomy at a single center between April and October 2012
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2012-10-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Correlation between early % total weight loss and % total weight loss 7 years following surgery. | A comparison made between 4 weeks and 7 years following the index surgery.
  A correlation between % total weight loss 4 weeks following surgery and % total weight loss at 7 years follow up based on clinic measurements.

SECONDARY OUTCOMES:
Reduction or cessation in the treatment for either type 2 diabetes mellitus and hypertension 7 years following surgery.. | A comparison was made between pre-operative medical / medication histories and equivalent data at 7 years follow up.
  Reduction / resolution of either hypertension or type 2 diabetes mellitus as defined by a reduction or cessation of medical treatment for the respective comorbidity. Patient diagnoses before surgery were compared with medical and medication histories taken at 7 years follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No